CLINICAL TRIAL: NCT07033845
Title: Pharmacokinetic Study of Topical Phenylephrine
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Daniel Alain, Inc. (Unknown); Follea International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DA-PK-001
Record Dates: First submitted 2025-05-22; First posted 2025-06-24 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Chemotherapy Induced Alopecia; Chemotherapy Side Effects
Keywords: Chemotherapy Induced Alopecia; Chemotherapy Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phenylephrine (Experimental): Topical Phenylephrine
  Interventions: Device: Phenylephrine

INTERVENTIONS:
Device: Phenylephrine — Topical Phenylephrine

SUMMARY:
Pharmacokinetic Study of Topical Phenylephrine

DETAILED DESCRIPTION:
A Phase 1 Open-Label Study to Evaluate the Pharmacokinetics of Topical Phenylephrine Applied to the Scalp in Healthy Adult Females

ELIGIBILITY:
Inclusion Criteria:

* Healthy females, age 18-55
* BMI: 18-30 kg/m²
* Fitzpatrick Skin Types I-IV (to standardize absorption risk)
* Scalp free from irritation, dermatologic disease, or damage
* Able to refrain from using other topical scalp products

Exclusion Criteria:

* History of cardiovascular disease, hypertension, or arrhythmia
* Scalp infections, wounds, or significant hair loss
* Recent use of medications that interfere with CYP enzymes or adrenergic systems
* Known sensitivity to phenylephrine or ethanol
* Positive drug screen or abnormal ECG at screening

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 24 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-10-19 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic profile of phenylephrine | Week [0,3]
  Determine the amount of phenylephrine and its metabolites in serum daily scalp application of topical phenylephrine for a period of 3 weeks

SECONDARY OUTCOMES:
Safety and tolerability of phenylephrine | Week [0, 3]
  Determine blood pressure and dermatological adverse events following daily scalp application of topical phenylephrine for a period of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andy Goren, MD, Study Director — University of Rome G. Marconi
Locations (1):
- University of Rome ("G. Marconi"), Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fahl WE. Complete prevention of radiation-induced dermatitis using topical adrenergic vasoconstrictors. Arch Dermatol Res. 2016 Dec;308(10):751-757. doi: 10.1007/s00403-016-1691-2. Epub 2016 Oct 4. PMID 27704205
- [Background] Soref CM, Fahl WE. A new strategy to prevent chemotherapy and radiotherapy-induced alopecia using topically applied vasoconstrictor. Int J Cancer. 2015 Jan 1;136(1):195-203. doi: 10.1002/ijc.28961. Epub 2014 May 16. PMID 24811525